CLINICAL TRIAL: NCT02109419
Title: Feasibility and Validity of A Novel Computer Based Battery For Analysis of Cognition, Mood, and Mobility-Independence in the Elderly
Brief Title: Feasibility and Validity of A Novel Computer Based Battery of Assessments in the Elderly
Acronym: HHT
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Corby K. Martin, Principal Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 2013-040
Record Dates: First submitted 2014-01-21; First posted 2014-04-09 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Computerized Assessment Feasibility and Validity
Keywords: computerized assessments; mood; cognition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All participants: All participants, including control, mild cognitive impairment, and dementia.
  Interventions: Other: HHT-G; Other: HHT-D; Other: Geriatric Depression Scale (DGS); Other: MMSE

INTERVENTIONS:
Other: HHT-G — Helping Hands Technology global cognitive function assessment
Other: HHT-D — Helping Hands Technology depression assessment
Other: Geriatric Depression Scale (DGS) — Geriatric Depression Scale (DGS)
Other: MMSE — Mini Mental State Exam

SUMMARY:
While standard pencil-and-paper test have continued to be useful for the monitoring of cognition, mood, and life space (LS) in the elderly they do have considerable limitations. Use of these pencil-and-paper tests requires that individuals come to the clinic for assessments, which results in significant clinical costs and practical limitations in the conducting of assessments in large numbers of individuals, and provides a time consuming and non-automated means of quantifying and recording changes in brain function. It is increasingly recognized that there is a need to develop valid and reliable computer based assessments to allow for the remote assessment of cognition, mood, and other parameters. Development of computerized based assessments will significantly increase the scale, scope, and speed with which cognition and mood can be measured in the elderly.

Helping Hands Technology LLC (HHT) has developed a number of web based assessments of cognition, mood, and LS. These new computerized assessments will be developed using new technology, and are based on the general principles found in existing pencil-and-paper based assessments of cognition, mood, and LS. In addition, HHT is developing proprietary means of reporting the results of the computerized assessments in an easy to use narrative format. This study will focus on quantifying the feasibility and validity of using HHT computerized assessments.

DETAILED DESCRIPTION:
See Brief Summary Section.

ELIGIBILITY:
Inclusion Criteria:

* Men and woman between the ages of 60-85, inclusive
* Cognitive function/impairment within appropriate ranges for the study (Mini-Mental State Exam scores of 10-30, inclusive)

Exclusion Criteria:

* Unable to complete computerized and standard pencil-and-paper based assessments

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will undergo screening to confirm eligibility, completion of initial screening form, and MMSE evaluation. Study subjects were enrolled with MMSE scores between 29-30, inclusive (healthy/control), 25-28, inclusive (mild cognitive impairment), and 10-24 (dementia).
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2014-03; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corby K Martin, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brouillette RM, Foil H, Fontenot S, Correro A, Allen R, Martin CK, Bruce-Keller AJ, Keller JN. Feasibility, reliability, and validity of a smartphone based application for the assessment of cognitive function in the elderly. PLoS One. 2013 Jun 11;8(6):e65925. doi: 10.1371/journal.pone.0065925. Print 2013. PMID 23776570
- [Background] Maerlender A, Flashman L, Kessler A, Kumbhani S, Greenwald R, Tosteson T, McAllister T. Examination of the construct validity of ImPACT computerized test, traditional, and experimental neuropsychological measures. Clin Neuropsychol. 2010 Nov;24(8):1309-25. doi: 10.1080/13854046.2010.516072. Epub 2010 Oct 4. PMID 20924979

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: All participants, including control, mild cognitive impairment (MCI), and dementia.
Period: Overall Study
Arm/Group | All Participants
Started | 57
Completed | 57
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants, inclusive of those with no memory impairment, mild cognitive impairment, and dementia.
Arm/Group | All Participants
Number analyzed (Participants) | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57
Geriatric Depression Scale (GDS) [Mean (Standard Deviation); unit: units on a scale] — Geriatric Depression Scale (GDS; min and max scores are 0 and 15, respectively; higher scores reflect higher depression).
  units on a scale | 1 (1.5)
Mini Mental State Questionnaire (MMSE) [Mean (Standard Deviation); unit: units on a scale] — Mini-Mental State Exam (MMSE; min and max scores are 0 and 30, higher scores reflect better cognitive functioning).
  units on a scale | 28 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Reliability and Validity of HHT's Computerized Assessments as Assessed by Correlation Analysis.
Description: Assess the reliability, validity and internal consistency of the HHT-D (Helping Hands Depression Test; min and max score is 0 and 30, respectively; higher scores reflect higher depression) and the HHT-G (Helping Hands global cognitive function screener; min and max scores are 0 and 30, respectively; higher scores reflect better cognition). In addition to assessing reliability, the HHT scales' validity was examined by correlating scores on the HHT scales with existing and already validated pen-and-paper assessments, which included the Mini-Mental State Exam (MMSE; min and max scores are 0 and 30, higher scores reflect better cognitive functioning), and the Geriatric Depression Scale (GDS; min and max scores are 0 and 15, respectively; higher scores reflect higher depression).
Time Frame: Visit completed over 16 day period
Population: Males and females between the ages of 60 and 85 years, inclusive, with MMSE scores of 10-30, inclusive.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- All Participants: All participants, including those with no memory impairment, mild cognitive impairment, and dementia.
Arm/Group | All Participants
Number analyzed (Participants) | 57
Units on a scale
  HHT-D Time 1/baseline | 11 (3.7)
  HHT-D Time 2, up to 16 days later | 11 (3.6)
  HHT-G Time 1/baseline | 25 (3.0)
  HHT-G Time 2, up to 16 days later | 25 (3.5)
Statistical Analysis 1: Comparison: All Participants; HHT-D reliability was evaluated via test-retest reliability coefficients. The dataset included participants from all groups; Test type: Other; p < 0.0001, Pearson Test-retest reliability coeff; Pearson Test-retest reliability coeff. = 0.80
Statistical Analysis 2: Comparison: All Participants; HHT-G reliability was evaluated via test-retest reliability coefficients. The dataset included participants from all groups; Test type: Other; p < 0.0001, Pearson test-retest reliability coeff; Pearson test-retest reliability coeff = 0.87
Statistical Analysis 3: Comparison: All Participants; Validity of the HHT-D was tested by Pearson correlation coefficients between HHT-D and Geriatric Depression Scale (GDS) scores. The dataset included participants from all groups; Test type: Other; p < .0001, Pearson correlation coefficient; Pearson correlation coefficient = 0.60
Statistical Analysis 4: Comparison: All Participants; Validity of the HHT-G was tested by Pearson correlation coefficients between HHT-G and Mini-Mental State Examination (MMSE) scores. The dataset included participants from all groups; Test type: Other; p = 0.0001, Pearson correlation coefficient; Pearson correlation coefficient = 0.71
Statistical Analysis 5: Comparison: All Participants; Internal consistency reliability of the HHT-D was assessed with Chronbach's alpha. The dataset included participants from all groups; Test type: Other; Chronbach's alpha = 0.73
Statistical Analysis 6: Comparison: All Participants; Internal consistency reliability of the HHT-G was assessed with Chronbach's alpha. The dataset included participants from all groups; Test type: Other; Chronbach's alpha = 0.70

ADVERSE EVENTS:
Groups:
- Control: Mini Mental State Exam (MMSE) score 29-30; inclusive
- Mild Cognitive Impairment: MMSE score 25-28; inclusive
- Dementia: MMSE score 10-24; inclusive
Arm/Group | Control | Mild Cognitive Impairment | Dementia
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24 | 0/8
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24 | 0/8

LIMITATIONS AND CAVEATS:
Test-retest reliability evaluated by administering the same battery at both time points in the study, hence learning effects were possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No